CLINICAL TRIAL: NCT01000181
Title: A Mechanistic, Non-randomised Study to Examine the Uptake of a Specific Radionuclide (61CuATSM) in Carotid Artery Plaque
Brief Title: Imaging 61CuATSM Uptake in Atherosclerotic Plaque Using PET-CT
Status: Suspended | Type: Observational
Why Stopped: Difficulty producing tracer
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Matthew Waltham, Senior Lecturer, King's College London
Other Study IDs: KCLADS09/1; GSTT Charity 251983; EudraCT 2009-011476-30
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases | interventions — CuATSM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing carotid endarterectomy
  Interventions: Other: PET-CT with CuATSM

INTERVENTIONS:
Other: PET-CT with CuATSM — PET-CT with CuATSM

SUMMARY:
The build up of plaque in the wall of the artery supplying blood to the brain poses a risk of stroke when the plaques become unstable and fragile. It is important to determine which patients are most at risk so that surgery can be performed. There is evidence that the risk is greatest when these plaques become oxygen deficient (hypoxic). The investigators wish to use PET imaging to identify hypoxic plaque, to help decide whether and when to perform surgery. The investigators have developed radiotracers (imaging agents) for this purpose, and this study is to determine whether they will work in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female patients who are 55yrs or older and for whom carotid endarterectomy is clinically indicated and a decision has been made to perform a carotid endarterectomy.
* Normal liver and adequate renal function. Assessed by measuring eGFR (>50ml/min) and creatinine (<130μmol/L)
* Life expectancy > 12 weeks
* Patients should be able to tolerate head/neck mask as well as lying in the PET-CT scanner

Exclusion Criteria:

* Abnormal liver and renal function (eGFR <50ml/min, Creatinine >130μmol/L)
* Patient unwilling to provide written informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-10

PRIMARY OUTCOMES:
Uptake of CuATSM in carotid plaque | Within 30 days of carotid endarterectomy

SECONDARY OUTCOMES:
Relationship of CuATSM uptake to plaque histology | Within 30 days of carotid endarterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Matt Waltham, MA PhD, Principal Investigator — King's College London
Locations (1):
- St Thomas' Hospital, London, United Kingdom